CLINICAL TRIAL: NCT04183036
Title: Endoscopic Sphincterotomy (EST) for Bile Duct Gallstones Cause Damage to the Ampulla of Vater and Sphincter of Oddi (SO): Endoclip Papillaplasty Help Recover the Damaged SO Function and Possibly Prevent Gallstone Recurrence
Brief Title: Endoclip Papillaplasty Recover Sphincter of Oddi Function After Endoscopic Sphincterotomy for Bile Duct Gallstones
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Huang Yonghui, chief physician, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: W201908
Record Dates: First submitted 2019-11-18; First posted 2019-12-03 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Sphincter of Oddi Function
Keywords: Choledocholithiasis; sphincterotomy;sphincter of Oddi
MeSH Terms: conditions — Choledocholithiasis

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Small EST combined with EPLBD (No Intervention)
- Large EST combined with ECPP (Experimental)
  Interventions: Procedure: Endoclip papillaplasty

INTERVENTIONS:
Procedure: Endoclip papillaplasty — Endoclip papilloplasty was performed to repair the Oddi sphincter using sterile repositionable hemostasis clipping device (Micro-tech (Nanjing), Co., Ltd.; stainless-steel). The operator positioned the clip and assessed the clip position and made sure the incision was clipped. Four to five endoclips were positioned in the incision in a zipper way from distal to proximal papillary sphincterotomy
  Arms: Large EST combined with ECPP

SUMMARY:
Gallstones in the common bile duct (CBD) may be asymptomatic but may lead to complications such as acute cholangitis or acute pancreatitis. EST is widely used for the treatment of bile duct gallstones. Despite its efficacy and improvements over time, EST is still associated with complications such as hemorrhage, perforation, pancreatitis, and permanent loss of function of the sphincter of Oddi (SO). Permanent loss of SO function can cause duodenobiliary reflux, bacterial colonization of the biliary tract, gallstone recurrence, cholangitis, and liver abscess.

Endoscopic papillary balloon dilation (EPBD) was first proposed in 1983 and it is now recognized as an alternative technique for the removal of CBD gallstones. The small balloon (diameter <8 mm) is less invasive, reduces the occurrence of adverse effects, and preserves the SO function, but it has limitations in the presence of CBD gallstones ≥10 mm in diameter. EST combined with endoscopic papillary large-balloon dilation (EPLBD) has been introduced for patients with large gallstone, but EPLBD widens the distal common bile duct and still may cause SO function damage, partially or completely. Repairing the ampulla of Vater and SO may reduce the long-term complication rates, especially gallstone recurrence. Unfortunately, no efficient strategy has been proposed. The present pilot study aimed to examine the feasibility and efficiency of an innovative strategy named endoclip papilloplasty to repair the damaged ampulla and recover SO function. The advantage of this device is that it can be rotated clockwise or counterclockwise by turning the handle until the correct position is achieved. Another advantage is if the clip is not in desired position, it may be re-opened and repositioned. Once satisfying clip positioning is achieved, the clip can be firmly attached to the tissue by pulling the slider back until tactile resistance is felt in the handle.Briefly, the operator assessed the patulous biliary opening and ductal axis, positioned and adjusted eachendoclip in order to close the patulous opening

DETAILED DESCRIPTION:
In order to reduce PEP risk, a rectal non-steroidal anti-inflammatory drug was administered 30 minutes before the ERCP in all patients. As the standard of care at the study hospital, the patients swallowed 2% lidocaine hydrochloride gel for local pharyngeal anesthesia, and 10 mg of diazepam were injected intramuscularly before ERCP. Anti-convulsants were not allowed. ERCP was performed in a standard manner using a side-viewing endoscope.

After successful selective deep cannulation of the common bile duct with a guidewire, the guidewire was extracted, and SOM was performed before contrast agent was introduced to determine the margins of the choledocholithiasis.

EST was performed, and the size of EST, which was large incision (incision to the full part of the ampulla) or long enough to ensure successful stone extraction, depended on the transverse diameter of the stones.

After stones removal, a 7.5Fr×26 cm biliary plastic stent, which was a suspended overlong biliary stent formed from a nasobiliary drainage tube (Boston Scientific), was placed to ensure that the biliary duct would not be clipped during endoclip papillaplasty and to reduce duodenobiliary reflux during the next 3-week before follow-up.

The investigators will recruit patients according to admission criteria and exclusion criteria. The participants underwent SOM before, immediately after EST, and 3 weeks after EST with endoclip papilloplasty. The participants were followed for 3 days during hospitalized. Complications including perforation, bleeding, and PEP were recorded. Blood routine, pancreatic enzymes (amylase and lipase), and liver function (serum alanine aminotransferase, aspartate aminotransferase, r-glutamyl transpeptidase, and alkaline phosphatase) were tested at 4 and 24 h after ERCP. All participants were followed at 3 weeks. The stent will be romoved with Allis clamp 3 weeks after the procedure.Symptoms were examined and blood tests as above were repeated ahead of stents retrieval and sphincter of Oddi monitoring through duodenoscope.

ELIGIBILITY:
Inclusion Criteria:

1)18-85 years of age; 2) informed consent obtained before ERCP; 3) CBD diameter ≥12 mm; 4) CBD gallstones visualized at magnetic resonance cholangiopancreatography (MRCP) with at least one gallstone ≥10 mm (transverse diameter)

Exclusion Criteria:

1. gallstone transverse diameter >35 mm, which is not appropriate to be extracted;
2. history of previous sphincterotomy, previous EPBD;
3. accompanied with choledochoduodenal fistula, coagulopathy, anticoagulant/antiplatelet therapy, or Billroth II or Roux-en-Y reconstruction;
4. papilla located deep within a diverticulum;
5. small papilla and short intramural segment, which was not suitable for large EST;
6. medications known to affect the SO (calcium channel blockers, nitrates, opiates, and anticholinergics) taken within 48 h of the procedure;
7. benign or malignant biliary stricture.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
SO manometric change | Before operation, During operation, Three weeks after operation
  The comparison of the SO manometric date before and after the procedure

SECONDARY OUTCOMES:
Frequency of use of ML and the incidence of adverse events | Three weeks after operation
  Mearsure the frequency of ML and the incidence of adverse events ，and to evaluate the healing of the ampulla

CONTACTS AND LOCATIONS:
Overall Officials: Yonghui Huang, MD, Principal Investigator — Peking University Third Hosptial
Locations (1):
- Xiue yan, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No